CLINICAL TRIAL: NCT00685126
Title: A Safety, Tolerability and Efficacy Study of Levalbuterol and Racemic Albuterol in Pediatric Subjects Birth to 48 Months Old With Reactive Airways Disease in an Acute Setting
Brief Title: Study of Levalbuterol and Racemic Albuterol in Pediatric Subjects With Reactive Airways Disease (RAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 051-033
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Reactive Airways Disease (RAD)
Keywords: RAD; Reactive Airways Disease; Levalbuterol; Racemic albuterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Low dose levalbuterol (0.15 mg, 0.31 mg or 0.63 mg); the first three doses will be delivered every 20 minutes for the first hour. Up to three additional doses may be given every 40 minutes thereafter. Additional doses may be administered at the investigator's discretion.
  Period II: Double blind, active-treatment period following discharge from the Emergency Department or Physician's Office. Subject will receive TID double-blind dosing. Period III: Double blind, active-treatment period following Visit 2. Subjects will receive double-blind dosing at the discretion of the investigator (PRN to TID).
  Interventions: Drug: Levalbuterol HCl Inhalation Solution
- B (Experimental): High dose levalbuterol (0.31 mg, 0.63 mg or 1.25 mg); the first three doses will be delivered every 20 minutes for the first hour. Up to three additional doses may be given every 40 minutes thereafter. Additional doses may be administered at the investigator's discretion.
  Period II: Double blind, active-treatment period following discharge from the Emergency Department or Physician's Office. Subject will receive TID double-blind dosing. Period III: Double blind, active-treatment period following Visit 2. Subjects will receive double-blind dosing at the discretion of the investigator (PRN to TID).
  Interventions: Drug: Levalbuterol HCl Inhalation Solution
- C (Active Comparator): Racemic albuterol (0.63, 1.25 mg or 2.5 mg); the first three doses will be delivered every 20 minutes for the first hour. Up to three additional doses may be given every 40 minutes thereafter. Additional doses may be administered at the investigator's discretion.
  Period II: Double blind, active-treatment period following discharge from the Emergency Department or Physician's Office. Subject will receive TID double-blind dosing. Period III: Double blind, active-treatment period following Visit 2. Subjects will receive double-blind dosing at the discretion of the investigator (PRN to TID).
  Interventions: Drug: Albuterol HCl Inhalation Solution

INTERVENTIONS:
Drug: Levalbuterol HCl Inhalation Solution — Nebulized unit dose vial for inhalation, low dose (0.15 mg, 0.31 mg or 0.63 mg), adjusted for body weight
  Other Names: Xopenex UDV; Xopenex Inhalation Solution; R-albuterol
  Arms: A
Drug: Levalbuterol HCl Inhalation Solution — Nebulized unit dose vial for inhalation, high dose (0.31 mg, 0.63 mg or 1.25 mg), adjusted for body weight
  Other Names: Xopenex UDV; Xopenex Inhalation Solution; R-albuterol
  Arms: B
Drug: Albuterol HCl Inhalation Solution — Nebulized unit dose vial for inhalation, dose (0.31 mg, 0.63 mg or 1.25 mg), adjusted for body weight
  Other Names: Ventolin; RS-albuterol
  Arms: C

SUMMARY:
The purpose of this study is to compare the efficacy of two dose levels of levalbuterol compared with one dose level of racemic albuterol in pediatric subjects aged birth to 48 months old.

DETAILED DESCRIPTION:
A double-blind, randomized, active-controlled, multicenter, parallel-group trial of levalbuterol in pediatric subjects presenting with acute reactive airways disease. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, must be between the ages of birth to 48 months inclusive at the time of consent.
* Subject must have experienced at least one previous episode or have a history of reactive airways disease.
* Subject must have an Oxygen saturation ≥ 90% at room air or with no more than 2 L/min supplemental Oxygen.

Exclusion Criteria:

* Subject who has participated in an investigational drug study within 30 days prior to study start, or who has previously participated in this study.
* Subject with a known sensitivity to levalbuterol or racemic albuterol, including Ventolin® or any of the excipients contained in any of these formulations.
* Subject using any prescription drug with which levalbuterol or racemic albuterol sulfate administration is contraindicated.

Max Age: 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2001-02; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Maximum decrease in Respiratory Status Scale© total score | Day 0: Approximately 5-10 minutes after each dose until subject is admitted or discharged

SECONDARY OUTCOMES:
Time to meet discharge criteria or clinical decision to discharge. | Days 0-7
Time to maximum decrease in Respiratory Status Scale© total score. | Days 0-7
Individual Respiratory Status Scale© items. | Days 0-7
Time to hospitalization. | Days 0-7
Rate of hospitalization. | Days 0-7

CONTACTS AND LOCATIONS:
Locations (34):
- United States (32):
  - Little Rock, Arkansas
  - Corona, California
  - Englewood, California
  - Huntington Beach, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Lake Worth, Florida
  - Tampa, Florida
  - Bloomington, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Marrero, Louisiana
  - Shreveport, Louisiana
  - Omaha, Nebraska
  - New York, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oswego, Ohio
  - Medford, Oregon
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Burke, Virginia
  - Norfolk, Virginia
  - Charleston, West Virginia
- Canada (2):
  - Halifax, Nova Scotia
  - Saskatoon, Saskatchewan